CLINICAL TRIAL: NCT05488860
Title: Piezoelectric Drived Microneedling in Treating Refractory Skin Diseases: A Pilot Study
Brief Title: Piezoelectric Drived Microneedling in Treating Refractory Skin Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XiangyaDerm0002
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Skin Diseases; Hypertrophic Scar; Keloid; Plantar Wart; Warts; Skin Tumor
Keywords: Microneedling; Ultrasound; Refractory skin diseases; Piezoelectric drived
MeSH Terms: conditions — Skin Diseases; Cicatrix, Hypertrophic; Keloid; Warts; Skin Neoplasms | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: Comparison is designed in each participant. For each individual, two similar hypertrophic scar/keloid or a single hypertrophic scar/keloid is randomly assigned into traditional injection group or piezoelectric divied microneedling group.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional injection (Active Comparator): Intralesional injection of drug by traditional injection needle. This is the traditional approach for drug delivery recommended by international guidelines for each skin diseases.
  Interventions: Drug: Triamcinolone acetonide(scar)/5-ALA(others)
- Piezoelectric drived microneedling (Experimental): Intralesional injection of drug by piezoelectric drived microneedles.
  Interventions: Procedure: Piezoelectric drived microneedling; Drug: 5-ALA (a photosensitizer for photodynamic therapy).

INTERVENTIONS:
Drug: Triamcinolone acetonide(scar)/5-ALA(others) — For scar, the drug is triamcinolone acetonide.
  Other Names: Intralesional drug delivery
  Arms: Traditional injection
Procedure: Piezoelectric drived microneedling — Piezoelectric drived microneedling
  Arms: Piezoelectric drived microneedling
Drug: 5-ALA (a photosensitizer for photodynamic therapy). — For other diseases, the drug is 5-ALA (a photosensitizer for photodynamic therapy).
  Arms: Piezoelectric drived microneedling

SUMMARY:
Piezoelectric drived microneedling treats refractory skin disorders using hollow microneedles assisted by ultrasound. Mechanically, the injection of medicine by hollow microneedling could makes the distribution of medicine more evenly. And the addition of ultrasound technique improves the effectiveness of microneedling. Investigators plan to conduct a pilot study to investigate the efficacy of using piezoelectric drived microneedles in treating refractory skin diseases.

DETAILED DESCRIPTION:
Piezoelectric drived microneedling treats refractory skin disorders using hollow microneedles assisted by ultrasound. Mechanically, the injection of medicine by hollow microneedling could makes the distribution of medicine more evenly. And the addition of ultrasound technique improves the effectiveness of microneedling. Investigators plan to conduct a pilot study to investigate the efficacy of using piezoelectric drived microneedles in treating refractory skin diseases. Investigators accept participants of hypertrophic scar, keloid and warts. For participants who are not candidates for traditional surgery, investigators will consider to accept carefully.

ELIGIBILITY:
Inclusion Criteria:

* Age over 16 years
* Diagnosed by 2 or more professional dermatologists
* Willing to underwent a new treatment modality
* Follow up is easy to conduct

Exclusion Criteria:

* Poor general condition
* Bleeding tendency
* Allergy to drug

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Short-term response | 1 week after treatment
  This is a qualitative item which should be evaluated by comparing the general images and dermoscopic images pre-treatment and post-treatment carefully.
Long-term response | 1 month after treatment
  This is a qualitative item which should be evaluated by comparing the general images and dermoscopic images pre-treatment and post-treatment carefully.

SECONDARY OUTCOMES:
Pain score during treatment | Immediately
  Using visual analogue scale (score 0-10, 0=no pain, 10=unbearable pain) to evaluate the level of pain
POSAS(The Patient and Observer Scar Assessment Scale) score | 1 month after treatment
  A widely used scar scale for evaluating the severity of scar by both patients and dermatologists. Score ranged from 11 to 110. The higher score means severer condition of scar.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, China

IPD SHARING:
Plan to Share IPD: No